CLINICAL TRIAL: NCT04145700
Title: A Randomized, Open-Label Phase 1/2 Study Evaluating Ramucirumab in Pediatric Patients and Young Adults With Relapsed, Recurrent, or Refractory Synovial Sarcoma
Brief Title: CAMPFIRE: A Study of Ramucirumab (LY3009806) in Children and Young Adults With Synovial Sarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated for meeting protocol specified futility criteria.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17306; J1S-MC-JV02 (Other: Eli Lilly and Company); 2018-004243-23 (EudraCT Number)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Synovial Sarcoma
Keywords: soft tissue sarcoma; adolescents and young adults (AYAs); adolescent
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma | interventions — Ramucirumab; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ramucirumab + Gemcitabine + Docetaxel (Experimental): Participants received intravenous (IV) infusions of ramucirumab 9 milligrams per kilogram (mg/kg), gemcitabine 900 milligrams per meter square (mg/m2) on days 1, 8, and docetaxel 75 mg/m2 on day 8 of a 21-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Ramucirumab; Drug: Gemcitabine; Drug: Docetaxel
- Gemcitabine + Docetaxel (Active Comparator): Participants received intravenous infusions of gemcitabine 900 mg/m2 on days 1, 8, and docetaxel 75 mg/m2 on day 8 of a 21-day cycle until disease progression or a criterion for discontinuation were met.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Ramucirumab — Ramucirumab given IV
  Other Names: LY3009806
  Arms: Ramucirumab + Gemcitabine + Docetaxel
Drug: Gemcitabine — Gemcitabine given IV
Drug: Docetaxel — Docetaxel given IV

SUMMARY:
This study is being conducted to test the safety and efficacy of ramucirumab in combination with other chemotherapy in the treatment of relapsed, recurrent, or refractory synovial sarcoma (SS) in children and young adults. This trial is part of the CAMPFIRE master protocol (NCT05999994) which is a platform to accelerate the development of new treatments for pediatric and young adult participants with cancer. Your participation in this trial could last 12 months or longer, depending on how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have discontinued all previous treatments for cancer or investigational agents ≥7 days after the last dose or per the type of previous treatment as stated in the protocol and must have recovered from the acute effects to ≤Grade 2 for alopecia and decreased tendon reflex and to ≤Grade 1 for all other effects at the time of enrollment, unless otherwise noted. Consult with the Lilly clinical research physician or scientist for the appropriate length of time prior to the first dose of study treatment.
* Participants with relapsed, recurrent, or refractory SS.
* Participants must:

  * Have measurable disease by Response Evaluation Criteria in Solid Tumors, Version (RECIST) 1.1.
  * have received at least one prior line of systemic treatment (including neoadjuvant and adjuvant chemotherapy) that contains ifosfamide and/or doxorubicin, or any approved therapies for which they are eligible, unless the patient is not a suitable candidate for the approved therapy.
  * not be eligible for surgical resection at time of enrollment.
* Adequate cardiac function, defined as: Shortening fraction of ≥27% by echocardiogram, or ejection fraction of ≥50% by gated radionuclide study.
* Adequate blood pressure (BP) control, defined as:

  * Participants ≥18 years: Controlled hypertension defined as systolic BP ≤150 millimeters of mercury (mmHg) or diastolic BP ≤90 mmHg where standard medical management is permitted. Please note that ≥2 serial BP readings should be obtained and averaged to determine baseline BP.
  * Participants <18 years: A BP ≤95th percentile for age, height, and gender measured as described in National High Blood Pressure Education Program Working Group (NHBPEPWG) on High Blood Pressure in Children and Adolescents (2004), where standard medical management is permitted. Please note that ≥2 serial BP readings should be obtained and averaged to determine baseline BP.
* Adequate hematologic function, as defined as:

  * Absolute neutrophil count (ANC): ≥750/microliters (µL) granulocyte-colony stimulating factor (G-CSF) permitted up to 48 hours prior. Participants with documented history of benign ethnic neutropenia or other conditions could be considered with a lower ANC after discussion with and approval from the Lilly clinical research physician or scientist.
  * Platelets: ≥75,000/cubic millimeters. Platelet transfusion permitted up to 72 hours prior.
  * Hemoglobin: ≥8 grams per deciliter (g/dL) (≥80 g/liter). Transfusions to increase the participant's hemoglobin level to at least 8 g/dL are permitted; however, study treatment must not begin until 7 days after the transfusion, and complete blood count criteria for eligibility are confirmed within 24 hr of first study dose.
* Adequate renal function, as defined as:

  * Creatinine clearance or radioscope glomerular filtration rate (GFR) ≥60 milliliters/minute/meters squared OR serum creatinine meeting the following parameters:

    * for participants ≥18 years of age serum creatinine ≤1.5×upper limit of normal (ULN);
    * for participants <18 years of age, serum creatinine based on age/gender as follows: Age 1 to <2 years maximum serum creatinine 0.6, Age 2 to <6 years maximum serum creatinine 0.8, Age 6 to <10 years maximum serum creatinine 1.0, Age 10 to <13 years maximum serum creatinine 1.2, Age 13 to <16 years maximum serum creatinine 1.5 for males and 1.4 for females, Age 16 to <18 years maximum serum creatinine 1.7 for males and 1.4 for females.
  * Urine protein meeting the following parameters:

    * for participants ≥18 years of age: <2+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <2 grams of protein in 24 hours to allow participation in the study.
    * for participants <18 years of age: ≤30 milligrams per deciliter urine analysis or <2+ on dipstick. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <1 g of protein in 24 hours to allow participation in the study.
* Adequate liver function:

  * Total bilirubin: ≤1.5×ULN. Except participants with document history of Gilbert Syndrome who must have a total bilirubin level of <3.0×ULN.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): ≤2.5×ULN OR ≤5.0×ULN if the liver has tumor involvement.
* The participant has an adequate coagulation function as defined by International Normalized Ratio ≤1.5 or prothrombin time ≤1.5×ULN, and partial thromboplastin time ≤1.5×ULN if not receiving anticoagulation therapy. For participants receiving anticoagulants, exceptions to these coagulation parameters are allowed if they are within the intended or expected range for their therapeutic use. Participants must have no history of clinically significant active bleeding (defined as within 14 days of first dose of study drug) or pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or known esophageal varices).
* The participant has adequate hematologic and organ function ≤1 week (7 days) prior to first dose of study drug.
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to randomization. Male and female participants must agree to use highly effective contraception for the duration of the study and up to 3 months following the last dose of ramucirumab and 6 months following the last dose of docetaxel and gemcitabine in order to prevent pregnancy.

Exclusion Criteria:

* Participants with severe and/or uncontrolled concurrent medical disease or psychiatric illness/social situation that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
* Participants who have active infections requiring therapy.

  * Participants with an active fungal, bacterial, and/or known severe viral infection including, but not limited to, human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).
* Participants who have had allogeneic bone marrow or solid organ transplant are excluded.
* Surgery: Participants who have had, or are planning to have, the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, or significant traumatic injury within 28 days prior to enrollment.
  * Central line placement or subcutaneous port placement is not considered major surgery.
  * Core biopsy, fine needle aspirate, and bone marrow biopsy/aspirate are not considered major surgeries.
  * Surgical or other wounds must be adequately healed prior to enrollment.
* Bleeding and thrombosis:

  * Participants with evidence of active bleeding or a history of significant (≥Grade 3) bleeding event within 3 months prior to enrollment are not eligible.
  * Participants with a bleeding diathesis or vasculitis are not eligible.
  * Participants with known or prior history in the prior 3 months of esophageal varices are not eligible.
  * Participants with a history of deep vein thrombosis requiring medical intervention (including pulmonary embolism) within 3 months prior to study enrollment are not eligible.
  * Participants with a history of hemoptysis or other signs of pulmonary hemorrhage within 3 months prior to study enrollment are not eligible.
* Cardiac:

  * Participants with a history of central nervous system (CNS) arterial/venous thromboembolic events (VTEs) including transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 6 months prior to study enrollment are not eligible.
  * Participants with myocardial infarction or unstable angina within the prior 6 months.
  * Participants with New York Heart Association Grade 2 or greater congestive heart failure (CHF).
  * Participants with serious and inadequately controlled cardiac arrhythmia.
  * Participants with significant vascular disease (eg, aortic aneurysm, history of aortic dissection).
  * Participants with clinically significant peripheral vascular disease.
* Participants who have a history of fistula, gastrointestinal (GI) ulcer or perforation, or intra-abdominal abscess within 3 months of study enrollment are not eligible.
* Participants with a history of hypertensive crisis or hypertensive encephalopathy within 6 months of study enrollment are not eligible.
* Participants who have non-healing wound, unhealed or incompletely healed fracture, or a compound (open) bone fracture at the time of enrollment are not eligible.
* Participants previously treated and progressed on combination gemcitabine and docetaxel regimen. Participants who received combination as maintenance therapy, without progression, would be eligible.
* Participants with a known hypersensitivity to ramucirumab, gemcitabine, docetaxel, or agents formulated with Polysorbate 80.
* Hepatic impairment:

  * Severe liver cirrhosis Child-Pugh Class B (or worse).
  * Cirrhosis with a history of hepatic encephalopathy.
  * Clinically meaningful ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
  * History of hepatorenal syndrome.
* The participant has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (eg, hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* The participant has symptomatic interstitial pneumonia or pulmonary fibrosis (or consistent findings of interstitial pneumonia/pulmonary fibrosis on imaging).
* Participants with central nervous system (CNS) involvement are ineligible.

Ages: 12 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (27):
  - Childrens Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Childrens Hospital of Orange County, Orange, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University Medical School, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Nationwide Children's Hosp, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Sydney Children's Hospitals Network, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Children's Hospital, Parkville, Victoria
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - UCL- Saint Luc, Brussels
- France (3):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Institut Curie, Paris
- Germany (3):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Italy (4):
  - Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Azienda Ospedaliera Di Padova, Padua
- Japan (2):
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Prinses Maxima Centrum, Utrecht
- Spain (5):
  - Hospital Universitario Virgen Del Rocio, Seville, Andalusia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
- United Kingdom (4):
  - The Christie, Manchester, Greater Manchester
  - University College Hospital - London, London
  - Royal Marsden Hospital, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: CAMPFIRE: A Study of Ramucirumab (LY3009806) in Children and Young Adults With Synovial Sarcoma — https://trials.lillytrialguide.com/en-US/trial/4Kdc8Gc0Rx6Z00sohuB8vD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completers included participants who died from any cause.
Groups:
- Ramucirumab + Gemcitabine + Docetaxel: Participants received intravenous infusions of ramucirumab 9 milligrams per kilogram (mg/kg), gemcitabine 900 milligrams per meter square (mg/m2) on days 1, 8, and docetaxel 75 mg/m2 on day 8 of a 21-day cycle until disease progression or a criterion for discontinuation were met.
Period: Overall Study
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
Started | 16 | 7
Received at Least One Dose of Study Drug | 16 | 6
Completed | 8 | 4
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ramucirumab + Gemcitabine + Docetaxel: Participants received intravenous infusions of ramucirumab 9 mg/kg, gemcitabine 900 mg/m2 on days 1, 8, and docetaxel 75 mg/m2 on day 8 of a 21-day cycle until disease progression or a criterion for discontinuation were met.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.70 (4.22) | 21.40 (4.58) | 18.80 (4.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 6 | 20
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 5 | 18
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 0 | 2 | 2
  Italy | 5 | 2 | 7
  Spain | 1 | 0 | 1
  United Kingdom | 6 | 2 | 8
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until the first investigator-determined objective progression as defined by Response Evaluation Criteria In Solid Tumors, Version 1.1 (RECIST v1.1) or death from any cause in the absence of progressive disease. Participants known to be alive and without disease progression will be censored at the time of the last adequate tumor assessment or date of randomization, whichever is later.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause (Up To 6.4 Months)
Population: All randomized participants (including the censored participants). Number of participants censored in Ramucirumab + Gemcitabine + Docetaxel=4, Gemcitabine + Docetaxel=2.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
Number analyzed (Participants) | 16 | 7
Months | 2.10 [2 to 6] | 2.03 [1.38 to NA] — There were not enough events to estimate the upper confidence limit.
Statistical Analysis 1: Comparison: Ramucirumab + Gemcitabine + Docetaxel vs Gemcitabine + Docetaxel; To conclude success for the intervention, the Bayesian analysis must yield a minimum of 99% posterior probability for PFS Hazard ratio less than 1 [i.e., Pr(HR < 1) > 99%]. The Bayesian analyses below include posterior mean of Hazard ratio, posterior probabilities instead of p-values, and credible intervals instead of confidence intervals; Test type: Superiority; p = 0.051, Bayesian hierarchical model; Posterior Mean Hazard Ratio = 2.62, 80% CI 2-sided [1.19 to 4.46]

2. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR)
Description: ORR is the best overall tumor response of complete response (CR) or partial response (PR) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up To 6.4 Months)
Population: All randomized participants.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
Number analyzed (Participants) | 16 | 7
Percentage of participants | 6.3 [0.7 to 22.2] | 0 [0 to 28]

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date that measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective disease progression is observed, per RECIST 1.1 criteria, or the date of death from any cause in the absence of documented disease progression or recurrence.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up To 4.13 Months)
Population: All randomized participants who had CR or PR responses. For Gemcitabine + Docetaxel, there were no participants with CR or PR responses to evaluate DoR, hence, zero participants analysed.
Measure: Number; unit: Months
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
Number analyzed (Participants) | 1 | 0
Months | NA — DoR couldn't be calculated as the participant did not achieve the event and was censored. |

4. Secondary Outcome: Complete Response (CR): Percentage of Participants Who Achieve CR
Description: CR is a disappearance of all target and non-target lesions and normalization of tumor marker level.
Time Frame: Baseline Up to 6.94 months
Population: All randomized participants.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
Number analyzed (Participants) | 16 | 7
Percentage of participants | 0 [0 to 13.4] | 0 [0 to 28]

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration of Ramucirumab (Cmax)
Description: Cmax was the concentration of study drug in the blood after the dose is administered. It was measured post-dose and was summarized using descriptive statistics.
Time Frame: 0.5 hours after the end of ramucirumab infusion on Day 1 of Cycle 1
Population: All randomized participants who received at least one dose of Ramucirumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 10
microgram per milliliter (µg/mL) | 231 (43)

6. Secondary Outcome: PK: Minimum Serum Concentration of Ramucirumab (Cmin)
Description: Cmin was the concentration of study drug in the blood immediately before the next dose was administered. It was measured pre-dose at all visits and was summarized using descriptive statistics.
Time Frame: Prior to ramucirumab infusion on Day 8 of Cycle 1, Day 1 of Cycle 2 and Day 1 of Cycle 5
Population: All randomized participants who received at least one dose of Ramucirumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel
Number analyzed (Participants) | 10
microgram per milliliter (µg/mL)
  Day 8 of Cycle 1: number analyzed (Participants) | 9
  Day 8 of Cycle 1 | 73.3 (39)
  Day 1 of Cycle 2 | 55.4 (24)
  Day 1 of Cycle 5: number analyzed (Participants) | 2
  Day 1 of Cycle 5 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there were only two participants. Individual values reported: 32.4 µg/mL, 41.3 µg/mL

7. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Drug Antibodies (TE-ADA)
Description: A TE-ADA evaluable participant is considered to be TE-ADA positive if the participant has at least one post baseline titer that is a 4-fold or greater increase in titer from baseline measurement (treatment-boosted). If baseline result is ADA Not Present, then the participant is TE ADA positive if there is at least one post baseline result of ADA Present with titer >= 20 (treatment-induced).
Time Frame: Baseline Up to 6.94 months
Population: All randomized participants who received at least one dose of study drug and had at least one non-missing baseline, post baseline ADA value.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
Number analyzed (Participants) | 7 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline Up to 6.94 months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Ramucirumab + Gemcitabine + Docetaxel | Gemcitabine + Docetaxel
All-Cause Mortality (participants affected / at risk) | 8/16 | 4/6
Serious Adverse Events (participants affected / at risk) | 8/16 | 2/6
Other Adverse Events (participants affected / at risk) | 15/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Gemcitabine + Docetaxel (N=16) | Gemcitabine + Docetaxel (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Gemcitabine + Docetaxel (N=16) | Gemcitabine + Docetaxel (N=6)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (11) | 1 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (11) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 2 (3)
Vomiting (Gastrointestinal disorders) | 7 (9) | 1 (3)
Asthenia (General disorders) | 2 (4) | 0 (0)
Fatigue (General disorders) | 4 (6) | 4 (5)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (9) | 0 (0)
Asymptomatic covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 2 (3) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (14) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 6 (10) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (10) | 0 (0)
Platelet count decreased (Investigations) | 6 (10) | 1 (4)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 4 (8) | 1 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatic nerve neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (9) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitation to this study was the highly varied estimates of the PFS HR and the probability of PFS HR < 1 due to influence from the matched historical controls whose PFS substantially outperformed PFS from the prospectively randomized control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT04145700/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04145700/SAP_001.pdf